CLINICAL TRIAL: NCT06055556
Title: Partial Heart Transplantation for Severe Pediatric Semilunar Valve Dysfunction
Brief Title: Partial Heart Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study no longer needed.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110600
Record Dates: First submitted 2023-08-23; First posted 2023-09-26 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partial Heart Transplantation (Experimental): Participants will receive a partial heart transplantation to replace the pulmonary valve with fresh donor graft(s). This is an investigational procedure. This means this procedure is not done as a routine treatment for patients with congenital heart defects. Partial heart transplantation involves surgical replacement of the semilunar heart valve with the heart valve and supporting blood vessels and tissue from an organ donor. No other parts of the heart are transplanted besides the heart valve, blood vessel, and tissue surrounding the valve.
  Interventions: Procedure: Partial Heart Transplantation; Other: Freshly procured valve

INTERVENTIONS:
Procedure: Partial Heart Transplantation — Partial heart transplantation involves surgical replacement of the semilunar heart valve with a fresh donor graft. The surgical procedure (homograft valve replacement) is common and standard of care. The investigational aspect of this is using a freshly procured valve rather than a cryopreserved, cadaveric one and also the use of limited immunosuppression to help maintain the freshly procured valve as "living tissue".
Other: Freshly procured valve — Fresh donor graft semilunar heart valve.

SUMMARY:
The purpose of this study is to determine if a partial heart transplantation in patients with congenital heart disease is safe and feasible. Participants will have a partial heart transplant involving surgical replacement of the pulmonary valve with the heart valve and supporting blood vessels from an organ donor. The procedure, tests, medications, and follow-up visits will all be done per standard of care. Medical data will be collected to look at outcomes after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a partial heart transplantation in patients with congenital heart disease is safe and feasible. Potential participants are patients 12 and younger with congenital heart defects in need of pulmonary valve replacement.Participants will have a partial heart transplant involving surgical replacement of the pulmonary valve with the heart valve and supporting blood vessels from an organ donor. The study procedure, tests, medications, and follow-up visits will all be done per standard of care for heart transplant patients. Data will be collected from chart review, before, during and after surgery and at standard of care follow-up visits. Study data will be compared to historical data of patients who have undergone other types of pulmonary valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart patient referred for a cardiac operation that involves valve replacement in pulmonary position
* Deemed acceptable for partial heart transplantation based on the standard evaluation process

Exclusion Criteria:

* Contraindication for heart transplantation
* Severe bliateral long segment pulmonary arterial hypoplasia
* Bilateral pulmonary vein stenosis
* Persistent acidosis with a pH < 7.1
* Failure to pass psychosocial evaluation
* Parental (custodial) alcohol and/or substance abuse
* Documented parental (custodial) child abuse or neglect
* Parent (custodian) with cognitive/psychiatric impairment severe enough to limit comprehension of medical regimen
* Infection disease exclusion criteria
* Evidence of active sepsis
* Hepatitis B surface antigenemia
* HIV positivity
* Pregnancy
* Financial hardship or insurance non-approval

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients who can be matched for transplant and the tissues needed procured | Day 1
  A measure of feasibility.
To assess valve growth following partial heart transplantation. | Year 2
  This will be determined by looking at valve growth compared to body growth over time based on post-operative imaging.

SECONDARY OUTCOMES:
To determine whether valve replacement(s) using partial heart transplantation is safe. | Year 2
  This will be determined by survival and major complication rates.
To assess valve function following partial heart transplantation. | Year 2
  This will be determined by looking for the development of valve stenosis over time based on post-operative imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Turek, MD, PhD, MBA, Principal Investigator — Duke Health
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No